CLINICAL TRIAL: NCT02892396
Title: Influence of Electronic Cigarettes in the Evaluation of the Inflammatory Response in Patients With a Diagnosis of COPD
Status: Completed | Type: Observational
Sponsor: Fundacio Catalana de Pneumologia (Other)
Responsible Party: Principal Investigator, Jacobo Sellarés Torres, Doctor in Medicine, Fundacio Catalana de Pneumologia
Other Study IDs: STUDY ECIGPOC
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood sample for study of inflammatory mediators.
  * Induced sputum culture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients & conventional cigarettes: COPD patients regular smokers of conventional cigarettes with no desire to quit smoking habit.
- COPD patients & electronic cigarettes: COPD patients who had been users of electronic cigarettes for at least 8 weeks. They will be provided with an specific type of electronic cigarette and the same dosage of inhaled nicotine.

SUMMARY:
This study evaluates the local and systemic inflammatory response in the airway in COPD patients who consume electronic cigarettes compared with conventional cigarette smokers.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is an illness with high morbidity and mortality in our society with a prevalence of about 10% of the population. Smoking represents the main risk factor for development of COPD having been associated with a greater decrease in lung capacity and increased mortality. Therefore, early treatment of smoking habit is an essential therapeutic approach.

The first line drug treatments have proven effective for smoking cessation, on the other hand the introduction of electronic cigarettes has brought a wide impact on our society,being considered as possible replacements in patients with difficulties in quitting the habit; however there is still limited information on its use in addition to some undesirable effects that have been described such as the lipoid pneumonia.

Recent clinical trials have shown that the use of electronic cigarettes may be associated with symptoms like dry cough, mouth irritation, dyspnea, and headache. On the other hand it has also been associated with increased airway resistance, an immediate decrease of exhaled nitric oxide (FeNO) and FEV1.

Our study aim to assess the inflammatory response in COPD patients who are regular consumers of electronic cigarettes compared with conventional cigarette smokers. The inclusion criteria in the study are: male patients diagnosed with COPD Gold B and C according to international guidelines that are regular smokers with no desire to quit their smoking habit. Exclusion criteria includes those with serious cardiovascular disease, chronic inflammatory disease, active oncologic disease of any origin, use of corticosteroids or other drugs with anti-inflammatory effect and finally COPD patients with acute exacerbation in the last twelve weeks.

Patients will be randomized into two groups: users of conventional and electronic cigarette. All patients in the second group will be provided with the same type of electronic cigarette and doses of inhaled nicotine.

We will perform a complete clinical characterization of the patients collecting data related with their smoking habit, daily consumption, tests to assess the degree of dependence and withdrawal symptoms, level of dyspnea and symptoms associated with tobacco consumption.

We will perform a complete respiratory functional test including spirometry, diffusion capacity and measurement of exhaled carbon monoxide levels. Inflammatory involvement of the airway will be examined by assessing the concentration of exhaled nitric oxide, studying the percentage of neutrophils and eosinophils in induced sputum and a general analysis for determination of inflammatory mediators: IL1B, IL6, IL8, factor alpha and C-reactive protein tumor necrosis.

The results will be evaluated by statistical tests. The results obtained will provide us with information about the effect of the electronic cigarette in COPD and its effectiveness in smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients Gold B or C
* Regular smokers with no desire to quit their habit.

Exclusion Criteria:

* Severe cardiovascular diseases.
* Chronic inflammatory diseases.
* Active oncologic diseases.
* Treatment with corticosteroids or other antiinflammatory drugs.
* Acute exacerbation of COPD in the last 12 weeks previous to their inclusion in the study

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male patients diagnosed with COPD Gold B or C according to international guidelines who have not had and acute exacerbation in the last 12 weeks prior to their inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of inflammatory response | 8 weeks
  Assessment of the local inflammatory airway response measured by respiratory functional test and sputum culture, in addition to the evaluation of the systemic inflammatory response provided by determination of acute reactants in blood tests (determination of C-reactive protein and cytokines in blood sample) in COPD patients.

SECONDARY OUTCOMES:
Clinical symptoms associated with COPD | 8 weeks
  Complete characterization of patients: tobacco consumption related symptoms: cough, oral irritation, dyspnoea. Control of the symptoms of nicotine withdrawal and evaluation test.
Tobacco withdrawal | 8 weeks
  Maintained smoking abstinence rate at 8 weeks in the electronic cigarette group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miravitlles M, Soriano JB, Garcia-Rio F, Munoz L, Duran-Tauleria E, Sanchez G, Sobradillo V, Ancochea J. Prevalence of COPD in Spain: impact of undiagnosed COPD on quality of life and daily life activities. Thorax. 2009 Oct;64(10):863-8. doi: 10.1136/thx.2009.115725. Epub 2009 Jun 23. PMID 19553233
- [Background] Sobradillo V, Miravitlles M, Jimenez CA, Gabriel R, Viejo JL, Masa JF, Fernandez-Fau L, Villasante C. [Epidemiological study of chronic obstructive pulmonary disease in Spain (IBERPOC): prevalence of chronic respiratory symptoms and airflow limitation]. Arch Bronconeumol. 1999 Apr;35(4):159-66. doi: 10.1016/s0300-2896(15)30272-6. Spanish. PMID 10330536
- [Background] Murray CJ, Lopez AD. Alternative projections of mortality and disability by cause 1990-2020: Global Burden of Disease Study. Lancet. 1997 May 24;349(9064):1498-504. doi: 10.1016/S0140-6736(96)07492-2. PMID 9167458
- [Background] Anthonisen NR, Connett JE, Murray RP. Smoking and lung function of Lung Health Study participants after 11 years. Am J Respir Crit Care Med. 2002 Sep 1;166(5):675-9. doi: 10.1164/rccm.2112096. PMID 12204864
- [Background] Anthonisen NR, Skeans MA, Wise RA, Manfreda J, Kanner RE, Connett JE; Lung Health Study Research Group. The effects of a smoking cessation intervention on 14.5-year mortality: a randomized clinical trial. Ann Intern Med. 2005 Feb 15;142(4):233-9. doi: 10.7326/0003-4819-142-4-200502150-00005. PMID 15710956
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Fairchild AL, Bayer R, Colgrove J. The renormalization of smoking? E-cigarettes and the tobacco "endgame". N Engl J Med. 2014 Jan 23;370(4):293-5. doi: 10.1056/NEJMp1313940. Epub 2013 Dec 18. No abstract available. PMID 24350902
- [Background] Abrams DB. Promise and peril of e-cigarettes: can disruptive technology make cigarettes obsolete? JAMA. 2014 Jan 8;311(2):135-6. doi: 10.1001/jama.2013.285347. No abstract available. PMID 24399548
- [Background] Caponnetto P, Campagna D, Cibella F, Morjaria JB, Caruso M, Russo C, Polosa R. EffiCiency and Safety of an eLectronic cigAreTte (ECLAT) as tobacco cigarettes substitute: a prospective 12-month randomized control design study. PLoS One. 2013 Jun 24;8(6):e66317. doi: 10.1371/journal.pone.0066317. Print 2013. PMID 23826093
- [Background] Vardavas CI, Anagnostopoulos N, Kougias M, Evangelopoulou V, Connolly GN, Behrakis PK. Short-term pulmonary effects of using an electronic cigarette: impact on respiratory flow resistance, impedance, and exhaled nitric oxide. Chest. 2012 Jun;141(6):1400-1406. doi: 10.1378/chest.11-2443. Epub 2011 Dec 22. PMID 22194587
- [Background] Hureaux J, Drouet M, Urban T. A case report of subacute bronchial toxicity induced by an electronic cigarette. Thorax. 2014 Jun;69(6):596-7. doi: 10.1136/thoraxjnl-2013-204767. Epub 2014 Jan 16. No abstract available. PMID 24436327
- [Background] McDonald VM, Higgins I, Wood LG, Gibson PG. Multidimensional assessment and tailored interventions for COPD: respiratory utopia or common sense? Thorax. 2013 Jul;68(7):691-4. doi: 10.1136/thoraxjnl-2012-202646. Epub 2013 Mar 16. PMID 23503624